CLINICAL TRIAL: NCT03928132
Title: Integrating Sex and Gender Considerations Into a Continuing Professional Development Activity on Diabetes and Depression: Protocol for a Non-Randomized Controlled Trial
Brief Title: Integrating Sex and Gender Into CPD for Depression/Diabetes
Acronym: INCluDED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Chaire Claire-Bonenfant-Femmes, Savoir et Société (Unknown); Institut du Savoir Montfort (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 384530
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Diabetes and depression; Continuing professional development; Continuing medical education; Sex and gender; Minority languages; Knowledge translation
MeSH Terms: conditions — Behavior; Diabetes Mellitus; Depression; Coitus

STUDY DESIGN:
Intervention Model Description: A non-randomized controlled trial
Who Masked: Participant
Masking Description: Health professionals will self-select their attendance at one or other of the interventions (control or experimental CPD activity) without knowing that they are different (one including sex and gender considerations, the other excluding them).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPD Workshop on Depression and Diabetes (Experimental): Participants in this arm will take part in a clinical CPD activity on depression and diabetes. The activity will include considerations of sex and gender, e.g. the different risk factors and impacts of treatment among women and men.
  Interventions: Behavioral: CPD Workshop on Depression and Diabetes
- CPD Workshop on Depression and Diabetes II (Sham Comparator): Participants in this arm will take part in a clinical CPD activity on depression and diabetes. The activity will exclude considerations of sex and gender, e.g. the different risk factors and impacts of treatment among women and men.
  Interventions: Behavioral: CPD Workshop on Depression and Diabetes

INTERVENTIONS:
Behavioral: CPD Workshop on Depression and Diabetes — 2 parallel face-to-face onsite workshops on diabetes and depression in primary care given by experts in French (control and experimental) using Powerpoint presentations.

SUMMARY:
People with type 2 diabetes are twice as likely to experience depression as nondiabetic individuals, and depression in turn increases the risk of diabetes. Clinical care for patients for either condition usually fails to consider the impact of sex and gender on tests, diagnosis and treatment, and evidence on these impacts is limited. The investigators aim to assess the impact of a continuing professional education activity (CPD) on diabetes and depression that includes considerations of sex and gender on the clinical behaviours of French-speaking healthcare professionals in Canada.

In a non-randomised controlled trial, the investigators are assessing the impacts of two CPD activities on depression and diabetes, one that includes considerations of sex and gender, and an identical one that omits sex and gender considerations, on French-speaking healthcare professionals' self-reported clinical behaviors regarding sex and gender considerations post-intervention and at 3 months. Data collection will occur in three distinct locations in Canada. Project development, data collection and analysis and dissemination of results will all integrate considerations of sex and gender. The process of creating a CPD activity that integrates considerations of sex and gender could be scaled up to other CPD activities in other clinical subjects and in other minority languages.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking health professionals (in practice and in training).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Immediate clinical behavioural intention, as measured by CPD-REACTION questionnaire | Immediately following the intervention
  Clinical behavioural intention to integrate considerations of sex and gender into the diagnosis and treatment of depression and diabetes, using the validated CPD-REACTION scale. CPD=continuing professional development, REACTION=a theoRy-basEd instrument to assess the impACT of continuing professional development activities on professional behavIOr chaNge. A 12-item Likert-type scale (i.e., Strongly disagree = 1, Strongly agree = 7; Never = 1, Always = 7, etc.) evaluates 5 constructs: 1) intention; 2) social influence; 3) beliefs about capabilities; 4) moral norms; and 5) beliefs about consequences. Sociodemographic questions are asked on sex, age (10 age ranges), province, rural/urban/semi-rural practice, and language of consultation. Mean, standard deviation, median and frequencies are calculated to summarize participant characteristics and questionnaire item responses. Construct scores are obtained by calculating the mean score for the items.
Change from immediate clinical behavioural intention at 3 months, as measured by CPD-REACTION questionnaire | 3 months after the intervention
  Evolution of clinical behavioural intention to integrate considerations of sex and gender into the diagnosis and treatment of depression and diabetes, using the validated CPD-REACTION scale, after a 3-month period.

SECONDARY OUTCOMES:
Acceptability Questionnaire | Immediately following the intervention.
  1) Participants rate acceptability of workshop with the following 9 items: organization, clarity, mastery of subject by trainer, exercises and discussion, presentation of sex and gender data, group interaction, overall quality, organization and quality of discussions and presentations, quality of documents distributed (Poor, Acceptable, Good, Very Good, or Excellent); 2) Participants rate the workshop length (too short, just right, too long); 3) Participants rate their confidence in incorporating the notions presented in the workshop in their management of Type 2 Diabetes (with or without depression) (scale of 1-10, 1=very little confidence, 10=very confident) both before and after the workshop; 4) Participants describe what changes they will make in their practice following the workshop; 5) Participants describe what they liked most and 6) least about the workshop; 7) Participants are asked if they thought the presentation was biased (yes/no) and if yes, are asked for details.

CONTACTS AND LOCATIONS:
Overall Officials: France Légaré, MD, PhD, Principal Investigator — CERSSPUL
Locations (1):
- CERSSPL, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate anonymous data only in the form of published results.

REFERENCES:
- [Derived] Deom Tardif A, Gogovor A, Guay-Belanger S, Audet D, Parent N, Gaudreau A, Remy-Lamarche D, Vigneault L, Ngueta G, Bilodeau A, Legare F; mATrICES-F Group. Integration of sex and gender in a continuing professional development course on diabetes and depression: a mixed methods feasibility study. BMJ Open. 2022 Apr 22;12(4):e050890. doi: 10.1136/bmjopen-2021-050890. PMID 35459660